CLINICAL TRIAL: NCT06604988
Title: Effectiveness of Video-feedback to Promote Positive Parenting in Families with Children At Risk of Autism Spectrum Disorder (ASD)
Brief Title: Effectiveness of Video-feedback for Positive Parenting with Children At Risk of ASD
Acronym: VIFEPOPA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Rosa Vilaseca, Associate professor, University of Barcelona
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 301104041962; PID2020-113401RB-I00 (Other Grant/Funding Number: Spanish Ministry of Economy and Competitiveness Fund)
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder (ASD; Parental Behaviors
Keywords: Parenting; Positive Parenting; Parental Behaviors; Adult-Child Interactions; Caregiver-Child Interaction; Autism Spectrum Disorder; Family intervention; Videofeedback intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Development of an evidence-based intervention to improve parenting. This evidence is based on a randomized controlled trial with longitudinal data collection. Once the informed consent is signed, all the information that will conform the baseline is collected (Wave 0) in all cases; those families meeting inclusion criteria will be provided with an alphanumeric label which corresponds to their anonymous identifier; families are then randomly assigned to the intervention or control groups according to a computer routine; during the following 6 months, measurements of some of the primary variables are collected up to a total of 3 times; after this time, the post-intervention measurement is collected (Wave 1); and finally a final collection is made after another 6 months (Wave 2).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A masking technique will be applied during the evaluation/recording phases of primary and secondary variables, as well as in the statistical analysis phase as described below. During the recording of variables, participants will only be identified by an alphanumeric label and without any reference to the group assigned at the beginning of the investigation. As regards data analysis, this will be carried out using anonymized databases and, automatically, a correspondence will be made between the participant&amp;#39;s identifier and the group to which he/she has been assigned to carry out the appropriate statistical analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group of videofeedback to promote positive parenting (Experimental): Biweekly sessions will be held for 6 months (a total of 12 sessions per family) via videoconference with the family at home. Each session will last approximately 1 hour to 1 hour and 30 minutes and will work with the primary caregiver. The intervention protocol mixes coaching strategies based on observation and video-feedback. This arm will provide with measurements at waves 0,1, and 2 over a time period of approximately 12 months.
  Interventions: Behavioral: Video-feedback intervention to promote positive parenting
- Control Group (No Intervention): This arm will only provide the measurements at the different time points (waves 0,1, and 2) over 12 months. After the follow-up planned in the study, feedback as well as recommendations concerning parenting will be provided.

INTERVENTIONS:
Behavioral: Video-feedback intervention to promote positive parenting — Each session will focus on three parental behaviours (that support child development) that have appeared clearly, frequently and consistently in the video (PICCOLO score of 2) in any of the 4 dimensions (affection, responsiveness, encouragement, teaching). Other aspects of parental behaviours that have scored 1 or 0 on the PICCOLO will also be considered, to increase their frequency or encourage their appearance. It is to be expected that all the behaviours collected in PICCOLO appear in one or more of the recordings, even if only occasionally. Behaviours that do not appear can be introduced through linking strategies with other behaviours in which parents show strength (for example, if a caregiver tends to name objects a lot, a link can be established between naming and asking the child the name of objects, if questions are behaviour that does not appear in the logs).
  In each session, the caregiver is shown video clips that clearly show the positive parenting behaviours.
  Arms: Intervention group of videofeedback to promote positive parenting

SUMMARY:
Improving parent-child interactions benefits child development and parents' perception of their competencies for childrearing and support for child learning and development, which in turns positively impacts on parental emotional well-being and Family Qualiy of Life.

This intervention protocol aims to improve the quality of parent-child interactions in daily-routine activities (bath time, dressing, mails…), specially during play interactions at home, increasing the frequency and consistency of the 29 positive parental behaviors included in the PICCOLO. PICCOLO is an observational tool for assessing positive parental behaviors in caregiver-child interactions that have been positively related to child cognitive, socioemotional, and linguistic development. It was developed and published in the United States, and it was validated in Spain with mothers and fathers. An Spanish handbook has been also published.

Guiding principles of the intervention protocol are an emphasis on the parents' strengths; a focus on daily routines in family context; and a non-directive intervention style, based on video feedback and coaching strategies as self-appraisal and reflection.

Although the protocol could be applied to different populations, this study is implemented with mothers and fathers with a young child (aged 24-36 months) at risk of Autism Spectrum Disorder (ASD). All children and their families are being cared for by professionals in Early Intervention Centers in Spain. Inclusion criteria for receiving this intervention are a) child at medium-high risk of ASD; b) primary caregiver at risk of anxiety, depression, or parental stress; c) primary caregiver with a low or medium-low level of positive parental behaviors in the PICCOLO.

The protocol includes bimonthly sessions of 60 minutes duration for six months with the main caregiver who participates in the program. Sessions are conducted by videoconference. Every session focuses on three different PICCOLO behaviors that have been identified in a previously recorded caregiver-child interaction during play at home (book-reading, symbolic play, or manipulative play). A new video is auto recorded every month by parents, so that each video is analyzed together with the caregiver in two sessions. After each session, the parents receive a written reminder of the aspects that have been worked on in the video feedback session, and of the agreements regarding the situations of daily life in which these aspects could be put into practice.

Family picture-books are progressively created, including selected frames from the videotapes that illustrate the positive parental behaviors that have been discussed. Six new images are included every month. Caregivers are encouraged to look at and talk about the book with their children at home and to share it with other family members.

The primary aim of the proposed study is to assess the efficacy of an intervention to improve caregiver competencies through the observation of caregiver-child interaction, using video-feedback coaching strategies based on parental strengths, from a collaborative model.

It is hypothesized that (1) developmentally supportive parental behaviors of mothers and fathers, measured with PICCOLO, after the intervention will be significantly higher in the intervention group (IG) than in the control group (CG); (2) levels of anxiety, or depression and/or stress of mothers and fathers after intervention will be significantly lower in the IG than in the CG; (3) Parental self-efficacy of mothers and fathers after the intervention will be significantly higher in the IG than in the CG; and (4) family quality of life after intervention will be significantly higher in the IG than in the CG. Also, it is hypothesized that individual trajectories in families within the IG will show changes in the outcome variables consistent with these expectations during the intervention period. it is hypothesized that these positive changes will not be observed in the CG, who will continue receiving the usual early intervention services.

With respect to intervention assessment, it is hypothesized that there will be significant and positive associations between key outcomes of the study and the scores obtained on the HOVRS-3 measure of four evidence-based home visiting practices: relationship building with families, responsiveness to family strengths, facilitating family interaction, collaboration with caregivers.

Finally, it is expected to find a secondary benefit on child's development, assessed with the DP-3 (Developmental Profile-3), particularly in the communication and social adaptation areas.

DETAILED DESCRIPTION:
The main objective of the study is to analyze the efficacy of a video feedback intervention in a group of mothers and fathers with children at risk of autism spectrum disorders (ASD). The intervention's impact on four variables will be assessed: parenting (1), the emotional distress of mothers and fathers (anxiety, depression and stress) (2), parental self-efficacy (3) and family quality of life (4). The differential change in individual trajectories will be analyzed for the four variables, based on belonging to the experimental group. The aim is to develop an intervention guide for the use of coaching strategies based on observation and video feedback.

Participants in the study will be 60 families comprised of a main caregiver (mother or father) of a child at risk of ASD between 24 and 36 months of age, with adequate internet access, who will be recruited from early intervention centers in Spain. The inclusion criteria are: a) the children have M-Chat scores compatible with medium-high risk of ASD (scores equal to or greater than 8); b) the main caregiver has high scores in at least one of the following variables: b.1) anxiety quantified using the HADS scale (scores equal to or greater than 7); b.2) depression quantified using the HADS scale (scores equal to or greater than 7); b.3) stress measured using the stress dimension of the PSI-F tool (scores equal to or greater than 86); c) the main caregiver has low parenting scores, quantified by the total score on the PICCOLO, an observational tool to score parental behaviors that support child development (score equal to or less than 40). The exclusion criteria are that the family: a) is currently receiving or has received in the last 12 months an intervention to improve parental interactions similar to the one proposed in this project or protocol; b) does not have a good level of written and spoken Spanish; or c) has mental health problems or children with serious physical problems or multiple disabilities.

The 60 families that meet the inclusion criteria will be randomly distributed into two groups of 30 families (intervention group and control group).

All the participants, both in the intervention group and the control group, will answer the questionnaires on emotional distress (anxiety, depression and parental stress), parental self-efficacy and family quality of life before and after the intervention. Child development will be evaluated before and after the intervention with the DP-3 instrument. Families will make an audiovisual recording of 10 minutes of play interaction at home with their child, under the conditions to which we will refer later.

For all the cases in the intervention group, the same protocol will be followed, which combines coaching strategies based on observation and video feedback.

Biweekly sessions will be conducted for 6 months (a total of 12 sessions per family) via videoconference with the family at home. Each session will last approximately between 1 hour and 1 hour 30 minutes and it will work with the main caregiver, following the following procedure.

Before the first session, the family is asked to record a 10-minute video of play interaction with their child at home in relation to three possible situations: i) reading books, ii) symbolic or fictional play, or iii) manipulative games (for example puzzles and shape fitting), using their own materials or games to be evaluated with PICCOLO. The analysis of this video recording assesses compliance with the inclusion criteria that refer to parental behaviors.

PICCOLO is an observational tool made up of 29 items that correspond to 29 developmental support parenting behaviors organized into four subscales or domains (affection, responsiveness, encouragement, teaching). The recording of a new video will be requested every two sessions, that is, at end of the evenly numbered sessions (2, 4, 6, etc.). Thus, each audiovisual record will be worked on during two sessions.

Before the first intervention session, a preliminary or reception session will be held. In this session, the first contact with the caregiver will be established to find out their concerns, interests and needs, to share with him/her what PICCOLO is (with an emphasis on positive parental behaviors and how these behaviors benefit and promote child development) and to explain the intervention procedure to the family. The main caregiver will be told that the focus of the intervention is positive parental behaviors observed in the videos and that in the sessions we will talk to the caregivers about these behaviors. The caregiver will be informed that in the first intervention session we will have seen the video that she sent us and we will focus on discussing some aspects of the interaction with her son or daughter. In the final part of this first reception session, the DP-3 development scale will be applied in an interview format (approximately 20 minutes), with the aim of collecting data about the child's development. It will be explained to the caregiver that collecting this information about the development of her son or daughter will help us to get to know him or her a little better. This scale of development is designed to be able to be applied virtually in an interview format with the main caregiver.

The procedure that will be followed in the other intervention sessions is as follows:

Each session will focus on three parental behaviors (that support child development) that have appeared clearly, frequently and consistently in the video (PICCOLO score of 2) in any of the 4 dimensions (affection, responsiveness, encouragement, teaching). Other aspects of parental behaviors that have scored 1 or 0 on the PICCOLO will also be taken into account, to increase their frequency or encourage their appearance. It is to be expected that all the behaviors collected in PICCOLO appear in one or more of the recordings, even if only occasionally. Behaviors that do not appear can be introduced through linking strategies with other behaviors in which parents show strength (for example, if a caregiver tends to name objects a lot, a link can be established between naming and asking the child the name of objects, if questions are behavior that does not appear in the logs).

In each session, the caregiver is shown video clips that clearly show the positive parenting behaviors and how they relate to what the child is doing, to give the primary caregiver the opportunity to observe themselves performing a positive parenting strategy or behavior. It is important to provide reflective feedback to caregivers. To give feedback to caregivers, we will choose three of the parenting behaviors and give the following message to parents:

"When I watched the video, I noticed that you [what the parent did], and that's [PICCOLO item label] in the [PICCOLO domain name] domain and I noticed [how the child responded] and that helps your child's development because [how it helps the child's development]. Let's talk about other times when you do these things and how you might be able to do them more often." Giving feedback with PICCOLO is simple if we plan our feedback focusing on three strong PICCOLO behaviours.

It is also important to give parents reflective feedback. We could use the following questions:

What do you think of this behaviour that we have been discussing? Had you noticed this? Do you think you could continue to do this? (Continue to ask questions based on the caregiver's responses and link them to the needs and/or concerns expressed by the family and to the child's development.

At what other times do you think you could do what we have discussed (family routines)?;How do you think you could do this? At the end of the session, we will close it with a brief summary of what was discussed and make an appointment for the next session.

At the end of the session, the intervener designs, in collaboration with the parents, an individualized biweekly family support programme (PIAFQ), in which they specify what other parental behaviours they can continue to carry out at home in their daily routines to promote the development of their children before the next intervention session.

The PIAFQ will be prepared in writing and sent to parents by email. In each session, the objectives of the previous fortnightly plan and how they have been carried out at home will be reviewed with the main caregiver. Doubts, needs and concerns of the caregiver will be addressed. These will vary for each child and family.

In addition, every two sessions the caregiver will be provided with visual support for the video feedback sessions in a book with pictures or images taken from the audiovisual records (electronic book, e-book, or a PowerPoint or PDF document).

Each page of the book will illustrate a parenting behavior that supports development and corresponds with an item of the PICCOLO. The image will be accompanied by a brief description of the parental behavior and its relationship with child development, in simple and direct language, as if the participants were speaking. You can include a footer (for example, "I love that my mom plays with me what I want to play" or "I like to encourage my son when he is struggling to fit the pieces in"), balloons typical of comics (for example, the mother says "I am happy when my daughter say a word or two and I can repeat what she says", "Yum, this soup is good!"). In addition, include some reference on the benefits for the child's development for example, "…and it helps me to learn words" or "…it makes me feel safe".

This picture book will be sent to parents along with the biweekly plan. Parents are encouraged to read the book with their child between video feedback visits, and to share it with other caregivers and/or family members of the child. This strategy has been used successfully in other studies to reinforce positive aspects of the interaction between the mother or the mother and her child. The intervention will be carried out by specialized professionals who are trained in video feedback by the main researchers of the project. Six months from the end of the intervention, follow-up measurements of all the study variables will be made in the intervention group and the control group.

ELIGIBILITY:
Inclusion Criteria:

Adequate family internet access. Child aged between 24 and 36 months. Child with a M-CHAT-R score compatible with high risk of ASD according to the manual (Score equal to or greater than 8 points).

Main caregiver with a high score in at least one of the following variables: a) anxiety quantified using the Hospital Anxiety and Depression Scale (HADS) (score equal to or greater than 7 points); b) depression quantified using the HADS (score equal to or greater than 7 points); c) stress measured using the stress dimension of the Parenting Stress Scale Short Form (PSI-F) (score equal to or greater than 86 points).

Main caregiver with a low level of developmentally supportive parental behaviors, quantified by the total score on the Spanish version of the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) (score equal to or less than 40 points). 40 points correspond to the 16% of the lowest scores in the Spanish validation sample for mothers, at 36 months of child's age.

Exclusion Criteria:

The family is currently receiving or has received in the last twelve months an intervention to improve parental interactions like the one proposed in this protocol, using positive feedback guidance based on observation of parent-child interaction.

Caregiver without a level of written and spoken Spanish that allows the intervention to be carried out.

Caregiver without internet connection for videoconferences. Caregiver with diagnosed mental health problems, excluding anxiety or depression symptoms.

Child with serious physical disability or multiple disabilities.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Parental anxiety | Pre-intervention, after six months of intervention, and follow-up six months later
  The Spanish version of the Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety symptoms in children's caregivers. The HADS is a self-reporting screening questionnaire composed of 14 items (seven items concerning depression symptoms and seven for anxiety symptoms) scored on a Likert scale from 0 to 3 points. Scores higher than 7 points in the subscale of anxiety symptoms, would indicate a risk of suffering health problems due to the mental issue assessed.
Parental depression | Pre-intervention, after six months of intervention, and follow-up six months later
  The Spanish version of the Hospital Anxiety and Depression Scale (HADS) will be used to assess depression symptoms in children's caregivers. The HADS is a self-reporting screening questionnaire composed of 14 items (seven items concerning depression symptoms and seven for anxiety symptoms) scored on a Likert scale from 0 to 3 points. Scores higher than 7 points in the subscale of depression symptoms, would indicate a risk of suffering health problems due to the mental issue assessed.
Parental stress | Pre-intervention, after six months of intervention, and follow-up six months later
  The Spanish version of the Parental Stress Scale (PSS) will be used to assess how caregivers perceive parental situations as stressful. This tool is composed of 12 items scored on a Likert scale, from 1 (total disagreement) to 5 (full agreement). The higher the score obtained, the higher the level of parental stress. Scores greater than or equal to 86 points would indicate a clinically significant parental stress score.
Parental behaviors ( Affection, Responsiveness, Encouragement, Teaching) | Pre-intervention, after six months of intervention, and follow-up six months later
  The Spanish version of the PICCOLO (Parenting Interactions with Children: Checklist of Observations Linked to Outcomes) will be used to assess parental behaviors. It is a reliable and validated 29-item measure of parent-child interactions for parents with children aged between 10 and 47 months old. The items are scored according to their frequency as 0 (absent, not observed), 1 (rare, minor or emerging) and 2 (clear, definitive, strong and frequent). The items are grouped into four domains: (a) Affection (7 items), which involves the physical and verbal expression of affection; (b) Responsiveness (7 items), which includes reacting sensitively to a child's cues and expressions; (c) Encouragement (7 items), which considers the parents' support of their child's efforts; and (d) Teaching (8 items), which includes cognitive stimulation, joint attention, and shared play. This tool has a total score between 0 and 58. Scores equal to or less than 40 points would indicate a low parenting score
Family Quality of Life | Pre-intervention, after six months of intervention, and follow-up six months later
  The Families in Early Intervention Quality of Life (FEIQoL) in its Spanish version will be used. The FEIQoL asks families to rate 39 FQoL features (i.e., items) on a 5-point rating scale from 1 = poor to 5 = excellent. The FEIQoL is comprised of four factors: family relationships, access to information and services, overall life situation, and child functioning. The minimum score on the scale is 39 points and the maximum score that can be obtained is 195 points. The higher the score obtained, the higher the level of Family Quality of Life. The scale shows a high internal consistency for the total score (α = .94) and its factors ranged from α = .74 to α = .89.
Parental self-efficacy | Pre-intervention, after six months of intervention, and follow-up six months later
  The Spanish version of the Parental Sense of Competence Scale (PSOC) will be administered to assess parental self-efficacy. The PSOC is a 17-item self-report scale that measures perceived parental self-efficacy. Responses are scored on a 6 point likert scale (from strongly disagree (1) to strongly agree (6)). The minimum score on the scale is 17 points and the maximum score that can be obtained is 102 points. Scores on the PSOC are transformed into three scores, a total score and a score for value/conforting dimension and the dimension of skills/conforting. The higher the score obtained, the higher the level of parental self-efficacy. The internal consistency coefficient was 0.85 for the total scale, and 0.78 and 0.85 for the two dimensions respectively.
Quality of intervention with caregivers | Intervention period
  To examine the quality of this highly individualized VFI process carried out with caregivers, four scales domains (relationship building with families, responsiveness to family strengths, facilitation of caregiver-child interaction, and collaboration with caregivers) of the Home Visit Rating Scale, version 3 (HOVRS-3) will be used.
  HOVRS-3 is structured in a list format, with each scale listing four to seven descriptive items, and each item followed by four quality indicators-1 (needs support), 3 (adequate), 5 (good), and 7 (excellent)-formatted similarly to multiple-choice test items. When the HOVRS-3 home-visit quality scores were higher, means a better quality of home visiting and it is related to parenting scores and children development. The scale demonstrated high values of validity and reliability (alphas between 0.69 to 0.91 depending on subscales) and adequate predictive validity.
Family satisfaction with the intervention | After six months of intervention
  To evaluate family satisfaction with the intervention, we will use the Spanish version of the Client Satisfaction Questionnaire (CSQ-8). It is a short questionnaire of 8 items with a likert-type response range from 1 to 4. It includes two open questions regarding the most valued aspects of the intervention and those that should be improved. The minimum score on the questionnaire is 8 points and the maximum score that can be obtained is 32 points. The higher the score obtained, the higher the level of satisfaction with the intervention. The original tool presented an adequate internal consistency, obtaining an alpha of 0.93. To add greater validity and to be able to obtain data on caregivers' perceptions of the quality of their working relationship with the VFI intervenor, we will use the Spanish version of the Working Alliance Inventory Adapted to Home Visiting - Short Revised (WAI -SR-HV).

SECONDARY OUTCOMES:
Children's development | Pre-intervention, after six months of intervention, and follow-up six months later
  The interview version of the Developmental Profile-3 (DP-3) will be used in the parent interview to assess child development. It consists of a total of 193 items that are not applied in their entirety in the interview version, but selected depending on the age of the boy or girl. It can be applied from birth to twelve years and eleven months of age. DP-3 is the Spanish adaptation of the latest version of the original Developmental Profile -II. Its constructs and theoretical structure are based on the multidimensional model of child development, which contemplates five major areas of development: motor skills, language and communication, socio-emotional development, cognitive development, and adaptive behavior. It is a screening test that allows a quick evaluation to detect possible delays in those five areas of child development, offering also a global development index of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Vilaseca, Psychology, Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon explicit request of the researchers to the Principal Researcher. We will have a longitudinal data collection. All participants meeting inclusion criteria will be provided with an alphanumeric label which corresponds to their anonymous identifier.
  The total scores for each variable and the aggregated data may be shared with explicit request to the Principal Investigator.

REFERENCES:
- [Background] Traube, D. E., Hsiao, H.-Y., Rau, A., Hunt-O'Brien, D., Lu, L., & Islam, N. (2020). "Advancing home based parenting programs through the use of telehealth technology": Correction. Journal of Child and Family Studies, 29(1), 54. https://doi.org/10.1007/s10826-019-01499-1
- [Background] Roggman L.A., Cook G.A., Innocenti M.S., Jump-Norman V. Parenting Interactions with Children: Checklist of Observations Linked to Outcomes: PICCOLO User's Guide. Paul, H. Brookes Publishing Co., Inc.; Baltimore, ML, USA: 2013. 92p
- [Background] Boyce, L.K., Innocenti, M.S., Roggman, L.A., Price, C., Jump V.K., Cook, G, & Ortiz, E. (2010). Family bookmaking: An approach to support parent-child language interactions in natural environments. Review of Disability Studies: An Inter-national Journal, 6, 42-53.
- [Background] Alpern, G. D. (2018). DP-3. Perfil de Desarrollo - 3 (F. Sánchez-Sánchez, adaptación española). Madrid: TEA Ediciones.
- [Background] Andrade-González, N., and Fernández-Liria, A. (2016). Spanish adaptation of the Working Alliance Inventory-Short (WAI-S). Current Psychology: A Journal for Diverse Perspectives on Diverse Psychological Issues, 35(1), 169-177. https://doi.org/10.1007/s12144-015-9365-3
- [Background] Gonzalez-Garcia RJ, Martinez-Rico G, Escorcia-Mora C, Garcia-Grau P. A Bibliometric Study on the Social Validity of Telepractice in Autism Spectrum Disorder. Int J Environ Res Public Health. 2022 Dec 27;20(1):419. doi: 10.3390/ijerph20010419. PMID 36612747
- [Background] Garcia-Grau P, Martinez-Rico G, Gonzalez-Garcia RJ, Escorcia-Mora CT, Canadas-Perez M. Caregiver Burden and Family Quality of Life in Early Intervention: The Role of Mothers and Family Confidence. Eur J Investig Health Psychol Educ. 2024 May 8;14(5):1325-1337. doi: 10.3390/ejihpe14050087. PMID 38785585
- [Background] Diaz-Herrero A, Lopez-Pina JA, Perez-Lopez J, Brito de la Nuez AG, Martinez-Fuentes MT. Validity of the Parenting Stress Index-Short Form in a sample of Spanish fathers. Span J Psychol. 2011 Nov;14(2):990-7. doi: 10.5209/rev_sjop.2011.v14.n2.44. PMID 22059342
- [Background] Vilaseca R, Rivero M, Bersabe RM, Cantero MJ, Navarro-Pardo E, Valls-Vidal C, Ferrer F. Demographic and Parental Factors Associated With Developmental Outcomes in Children With Intellectual Disabilities. Front Psychol. 2019 Apr 24;10:872. doi: 10.3389/fpsyg.2019.00872. eCollection 2019. PMID 31068864
- [Background] Vilaseca R, Rivero M, Ferrer F, Bersabe RM. Parenting behaviors of mothers and fathers of young children with intellectual disability evaluated in a natural context. PLoS One. 2020 Oct 13;15(10):e0240320. doi: 10.1371/journal.pone.0240320. eCollection 2020. PMID 33048940
- [Background] Roggman LA, Cook GA, Innocenti MS, Jump Norman VK, Boyce LK, Olson TL, Christiansen K, Peterson CA. The Home Visit Rating Scales: Revised, restructured, and revalidated. Infant Ment Health J. 2019 May;40(3):315-330. doi: 10.1002/imhj.21781. Epub 2019 Apr 1. PMID 30934132
- [Background] Walsh BA, Innocenti MS, Early S, Hughes-Belding K. Coaching home visitors: A thematic review with an emphasis on research and practice needs. Infant Ment Health J. 2022 Nov;43(6):959-974. doi: 10.1002/imhj.22016. Epub 2022 Oct 11. PMID 36219872
- [Background] Innocenti, M. S., Vilaseca, R., and Roggman, L. (2023). "PICCOLO: observing and coaching caregiver-child interaction to support early development in children with and without disabilities". in Family Centered Care in Childhood Disabil-ity. eds. L. Provenzi, S. Grumi, R. Borgatti, (Cham, CH: Springer) 115-147. doi: 10.1007/978-3-031-34252-3_7
- [Background] Rivero M, Vilaseca R, Cantero MJ, Valls-Vidal C, Leiva D. Relations between Positive Parenting Behavior during Play and Child Language Development at Early Ages. Children (Basel). 2023 Mar 3;10(3):505. doi: 10.3390/children10030505. PMID 36980063
- [Background] Roggman L.A., Cook G.A., Innocenti M.S., Jump Norman V., Christiansen K. Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PIC-COLO) in Diverse Ethnic Groups: PICCOLO Parenting Measure in a Diverse Sample. Infant Ment. Health J. 2013;34:290-306. doi: 10.1002/imhj.21389
- [Background] Vilaseca, R., Rivero, M., Leiva, D. et al. Mothers' and Fathers' Parenting and Other Family Context Variables Linked to Developmental Outcomes in Young Chil-dren With Intellectual Disability: A Two-wave Longitudinal Study. J Dev Phys Disabil 35, 387-416 (2023).
- [Background] Vilaseca R, Rivero M, Bersabe RM, Navarro-Pardo E, Cantero MJ, Ferrer F, Valls Vidal C, Innocenti MS, Roggman L. Spanish Validation of the PICCOLO (Parenting Interactions With Children: Checklist of Observations Linked to Outcomes). Front Psychol. 2019 Mar 27;10:680. doi: 10.3389/fpsyg.2019.00680. eCollection 2019. PMID 30971993
- [Derived] Vilaseca R, Rivero M, Leiva D, Roggman LA, Innocenti MS. The use of video feedback to promote developmentally supportive parent-child interactions with young children with ASD or at risk: study protocol for a randomized controlled trial (VIFEPOPA-RCT). BMC Psychol. 2025 Mar 4;13(1):196. doi: 10.1186/s40359-025-02494-6. PMID 40038736